CLINICAL TRIAL: NCT00890500
Title: A Phase I Study of Reduced Intensity, Sequential Double Umbilical Cord Blood Transplantation Using ProHema Modulated Umbilical Cord Blood Units in Subjects With Hematological Malignancies.
Brief Title: Safety and Efficacy of ProHema Modulated Umbilical Cord Blood Units in Subjects With Hematologic Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fate Therapeutics (Industry)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FT1050-01
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Hematologic Malignancies; Allogeneic Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Melphalan; Antilymphocyte Serum; Sirolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): 2 umbilical cord units: Second cord blood unit modulated with ProHema
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Antithymocyte Globulin; Drug: Sirolimus; Drug: Tacrolimus
- Group 2 (Active Comparator): 2 umbilical cord units: First cord blood unit modulated with ProHema
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Antithymocyte Globulin; Drug: Sirolimus; Drug: Tacrolimus

INTERVENTIONS:
Drug: Fludarabine — 30mg/m2/day IV x 6 days
Drug: Melphalan — 100 mg/m2/day IV x 1 day
Drug: Antithymocyte Globulin — 1mg/kg/day x 4 days
Drug: Sirolimus — GVHD Prophylaxis: Target range 3-12 ng/ml
Drug: Tacrolimus — GVHD Prophylaxis: Target range 5-10 ng/ml

SUMMARY:
The purpose of this research study is to determine the safety and efficacy of a reduced intensity conditioning regimen during a double umbilical cord blood unit transplant with one of the cord blood units modulated with ProHema.

DETAILED DESCRIPTION:
The purpose of this research study is to determine the safety and efficacy of a reduced intensity conditioning regimen during a double umbilical cord blood unit transplant with one of the cord blood units modulated with ProHema.

-As part of this research study cord units will be modulated in the laboratory with ProHema before it is given to the participant. Two different treatment groups will be tested. Group 1: will have the second cord blood unit modulated with ProHema; Group 2: will have the first cord blood unit modulated with ProHema.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies for whom allogeneic stem cell transplantation is deemed clinically appropriate
* Patient must be ineligible for traditional myeloablative transplantation according to treating physician
* Lack of 6/6 or 5/6 HLA-matched related, 8/8 HLA-matched unrelated donor, or unrelated donor not available within a time frame necessary to perform a potentially curative stem cell transplant
* 18-65 years of age
* ECOG Performance Status 0-2

Exclusion Criteria:

* The following hematologic malignancies are excluded:

  * Myelofibrosis unless there has been exposure to cytotoxic chemotherapy for the treatment of progression to acute myeloid leukemia
  * Chronic Myelogenous Leukemia, unless there has been exposure to cytotoxic chemotherapy for the treatment of blast phase, 3) Aplastic anemia, in the absence of transformation to Myelodysplastic disorder
* Cardiac disease: symptomatic congestive heart failure or evidence of left ventricular dysfunction as measured by gated radionucleotide ventriculogram or echocardiogram; active angina pectoris, or uncontrolled hypertension
* Pulmonary disease: symptomatic chronic obstructive lung disease, symptomatic restrictive lung disease, or corrected DLCO of < 50% of predicted, corrected hemoglobin
* Renal disease: serum creatinine > 2.0mg/dl
* Hepatic disease: serum bilirubin > 2.0mg/dl (expect in the case of Gilbert's syndrome or ongoing hemolytic anemia), SGOT or SGPT > 3 x upper limit of normal
* Neurologic disease: symptomatic leukoencephalopathy, active CNS malignancy or other neuropsychiatric abnormalities believed to preclude transplantation
* HIV antibody
* Uncontrolled infection
* Pregnancy or breast feeding mother
* Inability to comply with the requirements for care after allogeneic stem cell transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety of ProHema modulated umbilical cord blood units when used for transplantation in a reduced intensity, sequential umbilical cord blood transplantation model. | 2 years

SECONDARY OUTCOMES:
Time to engraftment of umbilical cord blood units | 2 years
Fractional chimerism of transplanted cord blood units | 2 years
Rates of acute and chronic GVHD | 2 years
30- and 100-day treatment related mortality | 2 years
Measures of immune reconstitution and relapse-free and overall survival at 1 and 2 years after transplantation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Corey Cutler, MD, MPH, FRCP(C), Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Cutler C, Multani P, Robbins D, Kim HT, Le T, Hoggatt J, Pelus LM, Desponts C, Chen YB, Rezner B, Armand P, Koreth J, Glotzbecker B, Ho VT, Alyea E, Isom M, Kao G, Armant M, Silberstein L, Hu P, Soiffer RJ, Scadden DT, Ritz J, Goessling W, North TE, Mendlein J, Ballen K, Zon LI, Antin JH, Shoemaker DD. Prostaglandin-modulated umbilical cord blood hematopoietic stem cell transplantation. Blood. 2013 Oct 24;122(17):3074-81. doi: 10.1182/blood-2013-05-503177. Epub 2013 Aug 30. PMID 23996087